CLINICAL TRIAL: NCT01960283
Title: Randomized Clinical Trial Evaluating the Efficacy of Methotrexate in Addition to Anti-H1 Versus Placebo and Anti-H1 in the Treatment of Severe Chronic Idiopathic Urticaria
Brief Title: Methotrexate in the Treatment of Chronic Idiopathic Urticaria
Acronym: MUCIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRN09-AM/MUCIS
Record Dates: First submitted 2013-01-15; First posted 2013-10-10 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Active Comparator): The group I will receive the intervention :
  Methotrexate + anti-H1
  Interventions: Drug: Methotrexate (Novatrex ®) + anti-H1
- Group II (Placebo Comparator): The intervention in group II will include : placebo + anti-H1
  Interventions: Drug: Placebo + anti-H1

INTERVENTIONS:
Drug: Methotrexate (Novatrex ®) + anti-H1 — Methotrexate (Novatrex ®) tablets 2.5 mg methotrexate 0.2 mg/kg/week as a single dose, orally for 8 weeks.
  After 8 weeks, if the treatment is still not efficient, the dose will be increased to 0.25 mg/kg/week and continued until W18.
  For anti-H1 treatment, the same molecules with the same dosage than before the recruitment will be continued, and methotrexate will be added in this group.
  Other Names: Methotrexate; Anti-H1
  Arms: Group I
Drug: Placebo + anti-H1 — Placebo: 0.2 mg / kg / week as a single dose, orally for 8 weeks. After eight weeks, if the patient is still very embarrassed, the dose is increased to 0.25 mg / kg / week in a weekly dose.
  For anti-H1 treatment, the same molecules with the same dosage than before the recruitment will be continued, and the placebo of methotrexate will be added in this group.
  Other Names: Placebo of methetrexate + anti-H1
  Arms: Group II

SUMMARY:
Chronic urticaria is defined by urticarial lesions persisting at 6 weeks. The cause is not found in about 75% of cases (chronic idiopathic urticaria). The gold standard treatment consists of anti-H1 molecules. In severe cases, refractory to anti-H1, few therapeutic alternatives exist. Methotrexate, which is not expensive and often prescribed by dermatologists, has been efficiently tried in an open study on severe chronic idiopathic urticaria, and also in few case reports.

DETAILED DESCRIPTION:
Chronic urticaria, defined by its persistence beyond 6 weeks, is a common condition (0.1% to 3% of the general population), occurring at any age. The etiology is not found in nearly 75% of cases (chronic idiopathic urticaria). Chronic idiopathic urticaria may resolve over several months or years. The quality of life of patients is usually strongly spoiled. The gold standard treatment consist of anti-H1 molecules. In severe cases, which are refractory to anti-H1, few therapeutic alternatives exist. Two studies have shown a benefit when adding to anti-H1, montelukast, anti-leukotriene, or cyclosporine. Methotrexate, which is another immunosuppressive drug, cheap and commonly prescribed by dermatologists, has been efficient in severe chronic urticaria, in an open study and in few case reports.

Methotrexate, an anti-metabolite drug which inhibits dihydrofolate reductase, is indicated in hematologic malignancies and in autoimmune diseases. It may be given by oral or parenteral administration, once a week, and requires regular monitoring of renal and hepatic function, and blood count.

ELIGIBILITY:
Inclusion Criteria:

Patients who met the diagnostic criteria for chronic idiopathic urticaria, previously treated by

* 3 different molecules of anti-H1 or
* a combination of 2 different molecules of anti-H1 or
* 1 molecule of anti-H1 with at least a double dose for a total treatment duration of ≥ 3 months before inclusion
* With persistency of at least 7 days with urticarial lesions in the previous month

Exclusion Criteria:

* Differential diagnosis of chronic idiopathic urticaria (urticarial vasculitis)
* Treatment with montelukast or immunosuppressive drugs during the previous month
* Contraindications to methotrexate

  * Allergy to methotrexate
  * Treatment which are contraindicated with methotrexate
  * Pregnancy, possibility of getting pregnant (no effective contraception), breastfeeding
  * Anomalies in liver function (transaminases or liver failure at a rate 1.5 X normal)
  * Severe renal impairment (creatinine clearance calculated by the cockcroft formula <50 ml / min)
  * Chronic respiratory failure
  * Active infectious chronic diseases (viral hepatitis, HIV)
  * History of neoplasia
  * Mental deficiency
  * Involvement in another drug clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete remission of urticaria at 18 weeks | at 18 weeks of treatment
  Number of patients with complete remission of urticaria at 18 weeks, defined as no urticarial lesion 30 days before W18

SECONDARY OUTCOMES:
Tolerance : clinical and biological safety | 18 weeks
  Number of patients with clinical adverse effects Number of patients with biological adverse effects
Efficacy of the treatment in improving symptoms : pruritus | 18 weeks and 26 weeks
  Number of patients with :
  - pruritus At 18 weeks and 26 weeks
Persistency of the complete remission at 26 weeks | 26 weeks
  Number of patients with persistency of the complete remission, defined as no urticarial lesion from the withdrawal of treatment until W26
Efficacy of the treatment in improving symptoms : outbreaks by week | 18 weeks and 26 weeks
  - number of outbreaks by week/patient At 18 weeks and 26 weeks
Efficacy of the treatment in improving symptoms : duration of lesions | 18 weeks and 26 weeks
  - mean +/- standard deviation duration of lesions At 18 weeks and 26 weeks
Efficacy of the treatment in improving quality of life | 18 weeks and 26 weeks
  Mean DLQI (quality of life) score :
  At 18 weeks and 26 weeks
Efficacy of the treatment in improving quality of sleep | 18 weeks and 26 weeks
  Mean score of quality of sleep (from 0 to 100) At 18 weeks and 26 weeks
Efficacy of the treatment in improving facial/cervical urticarial lesions | 18 weeks and 26 weeks
  Number of patients with, either :
  * facial/cervical urticarial lesions
  * urticarial lesions on the body only
  * facial/cervical + body lesions Indeed, facial or cervical urticarial lesions are considered more disturbing. At W18 and W26

CONTACTS AND LOCATIONS:
Overall Officials: Annabel MARUANI, MD, PhD, Principal Investigator — University Hospital of Tours, France
Locations (11):
- France (11):
  - CHRU BREST Morvan, Brest
  - Chu Mondor, Créteil
  - Ch Le Mans, Le Mans
  - CHRU LILLE Huriez, Lille
  - CHRU NANCY Brabois, Nancy
  - Chru Nantes, Nantes
  - Hopital TENON, Paris
  - CHRU POITIERS La Miléterie, Poitiers
  - Chru Reims, Reims
  - CHRU RENNES Pontchaillou, Rennes
  - Chru Tours, Tours